CLINICAL TRIAL: NCT06938581
Title: The Utility of Enhanced Recovery After Surgery (ERAS) Protocols in Breast Conserving Surgery: A Randomized Control Trial
Brief Title: ERAS Protocols in Breast Conserving Surgery
Acronym: ERAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0132-25-FB
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Postoperative Recovery
Keywords: Eras; Opioid Use; Pain Management; Breast Conserving Surgery; Sentinel Lymph Node Biopsy; Perioperative Care
MeSH Terms: conditions — Breast Neoplasms; Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ERAS Protocol Arm (Active Comparator): Participants will receive the Enhanced Recovery After Surgery (ERAS) protocol as part of peri-operative care. The ERAS protocol includes: (day before surgery) oral carbohydrate drink in the evening, Acetaminophen 1000mg in the evening, Celecoxib 200mg in the morning and evening and (morning of surgery) oral carbohydrate drink 2-4 hours before surgery, Celecoxib 200mg, Acetaminophen 1000mg.
  Additionally, peri-operative medications such as Acetaminophen, Scopolamine, Dexamethasone, and Ondansetron may be given as needed at the discretion of the surgery and anesthesia teams.
  Interventions: Other: ERAS Protocol
- Standard Care Arm (Experimental): Participants will receive standard peri-operative care without the Enhanced Recovery After Surgery (ERAS) protocol. This includes routine preoperative instructions and omission of the ERAS-specific interventions (oral carbohydrate drink, Celecoxib, and preoperative Acetaminophen). Perioperative medications such as Acetaminophen, Scopolamine, Dexamethasone, and Ondansetron may be given as needed at the discretion of the surgery and anesthesia teams.
  Interventions: Other: Standard Perioperative Care

INTERVENTIONS:
Other: ERAS Protocol — The ERAS protocol consists of:
  * Day before surgery: Oral carbohydrate drink (evening), Acetaminophen 1000mg (evening), Celecoxib 200mg (morning and evening)
  * Morning of surgery: Oral carbohydrate drink (2-4 hours before surgery), Celecoxib 200mg, Acetaminophen 1000mg Additionally, optional perioperative medications (Acetaminophen, Scopolamine, Dexamethasone, Ondansetron) may be given as needed.
  Arms: ERAS Protocol Arm
Other: Standard Perioperative Care — Standard perioperative care without ERAS protocol components. Includes routine preoperative instructions and omission of oral carbohydrate drink, celecoxib, and preoperative acetaminophen. Optional perioperative medications (Acetaminophen, Scopolamine, Dexamethasone, Ondansetron) may be given as needed.
  Arms: Standard Care Arm

SUMMARY:
Enhanced Recovery After Surgery (ERAS) protocols have been of increasing interest in the surgical community for decades. The emphasis has been development of protocols to maximize pain control post-operatively without the use of opioids. While this approach has been studied extensively in the oncology surgery literature, little data exists on the utility of ERAS protocols in the setting of breast conserving surgery (BCS), which is a type of surgery to remove breast cancer while saving as much of the breast as possible. The purpose of this study is to determine the utility of implementing ERAS protocols in breast cancer patients undergoing breast conserving surgery. Study participants will be randomized to either ERAS protocol or standard peri-operative care without ERAS. The study will assess the how many opioid prescriptions are given in the first week after surgery and how much pain participants report right after surgery. Investigators will also look at how long participants stay in the recovery room and if medicine for nausea is needed.

DETAILED DESCRIPTION:
Enhanced Recovery After Surgery (ERAS) protocols have been of increasing interest in the surgical community for decades. The emphasis has been development of protocols to maximize pain control post-operatively without the use of opioids. While this approach has been studied extensively in the oncology surgery literature, little data exists on the utility of ERAS protocols in the setting of breast conserving surgery (BCS). The study aims to enroll 260 participants undergoing breast conserving surgery (lumpectomy with sentinel lymph node biopsy) for cT1-T3 N0 breast cancer. Participants will be randomly assigned to either the ERAS protocol or standard peri-operative care without ERAS.

The ERAS protocol is comprised of celecoxib 200mg, morning and evening, and an oral carbohydrate drink and acetaminophen 1000mg in the evening the day before surgery and an oral carbohydrate drink (2-4 hours before surgery), celecoxib 200mg and acetaminophen 1000mg the morning of surgery. Participants in the standard care arm will receive routine peri-operative instructions without ERAS interventions. The study's primary objectives are to determine the proportion of participants receiving an opioid prescription within 7 days after surgery and to evaluate the participant-reported pain levels in the post-anesthesia care unit (PACU) using the Numerical Rating Scale (NRS). The secondary objectives are to determine the length of stay in PACU and the use of anti-emetic medications in PACU. The study uses a non-inferiority design to test if standard care without ERAS is not significantly worse than ERAS for opioid use and pain scores. Statistical comparisons will look at proportions and averages between the ERAS and standard care groups, with additional analysis based on tumor size.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 19 years of age or older
* Able to provide study-specific informed consent
* Histologic confirmation of breast cancer on core needle biopsy
* Clinical or radiographic cT1-T3 N0 disease
* Undergoing breast conserving surgery with lumpectomy & sentinel lymph node biopsy
* No prior definitive treatment or intervention
* Able to swallow and retain oral carbohydrate drinks and medication

Exclusion Criteria:

* Pregnant
* Contraindications to ERAS protocol components
* Undergoing lumpectomy without sentinel lymph node biopsy, mastectomy, or other specified procedures
* Diagnosed with cT4 or N1-3 disease
* Metastatic disease at presentation
* Taking opioid pain medications for other indications
* History of substance use disorder
* Any condition where ERAS could compromise safety

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants With Opioid Prescriptions Within 7 Days of Surgery | Within 7 days post-surgery
  The percentage of participants who receive an opioid prescription from the surgery team within 7 days after surgery will be determined from the documented electronic medical record.
Immediate Post-operative Pain Score | Within 24 hours post-surgery
  Participant reported pain level in the post-anesthesia care unit (PACU) using the Numerical Rating Scale (NRS) will be assessed. Scoring is from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Post-anesthesia Care Unit Length of Stay | Within 48 hours post-surgery
  The duration of time in minutes from arrival in the post-anesthesia care unit (PACU) to discharge home will be recorded.
Use of Anti-emetic Medication in Post-anesthesia Care Unit | Within 48 hours post-surgery
  The proportion of participants who receive any anti-emetic medication (such as ondansetron, prochlorperazine, haloperidol, or metoclopramide) from arrival in the PACU to discharge home will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Santamaria, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cyr AE. Underutilization of Enhanced Recovery After Surgery (ERAS) in Breast Surgery: An Opportunity to Reduce Opioid Usage. Ann Surg Oncol. 2020 Apr;27(4):966-968. doi: 10.1245/s10434-020-08198-y. Epub 2020 Jan 23. No abstract available. PMID 31974707
- [Background] Chiu C, Aleshi P, Esserman LJ, Inglis-Arkell C, Yap E, Whitlock EL, Harbell MW. Improved analgesia and reduced post-operative nausea and vomiting after implementation of an enhanced recovery after surgery (ERAS) pathway for total mastectomy. BMC Anesthesiol. 2018 Apr 16;18(1):41. doi: 10.1186/s12871-018-0505-9. PMID 29661153
- [Background] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Background] Batdorf NJ, Lemaine V, Lovely JK, Ballman KV, Goede WJ, Martinez-Jorge J, Booth-Kowalczyk AL, Grubbs PL, Bungum LD, Saint-Cyr M. Enhanced recovery after surgery in microvascular breast reconstruction. J Plast Reconstr Aesthet Surg. 2015 Mar;68(3):395-402. doi: 10.1016/j.bjps.2014.11.014. Epub 2014 Nov 21. PMID 25488326